CLINICAL TRIAL: NCT06623006
Title: Self Management of Type 2 Diabetes Using a Co-designed Mobile Health (mhealth) Intervention in Nepal: a Randomized Control Trial
Brief Title: Self Management of Type 2 Diabetes Using a Text Based Mobile Health (mhealth) Intervention in Nepal
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Huddersfield (Other)
Responsible Party: Principal Investigator, Namuna Shrestha, PhD student-full time, University of Huddersfield
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: UHuddersfieldProtV000001
Record Dates: First submitted 2024-09-30; First posted 2024-10-02 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-09

CONDITIONS: Type 2 Diabetes Mellitus (T2DM)
Keywords: type 2 diabetes, mhealth, self-management, Nepal
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Telemedicine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control group (No Intervention): The control group will be receive usual care they have been getting. At the end of the intervention, they will be provided with a leaflet that contains messages that was included in the mhealth intervention.
- Intervention (Experimental): The intervention group will receive a text-based mhealth (text messages) in addition to standard care which they are used to receiving.
  Interventions: Behavioral: mobile health (mhealth)

INTERVENTIONS:
Behavioral: mobile health (mhealth) — The intervention will include a text-based mhealth component, designed using a behaviour change framework (Behaviour Change Wheel). The development process will be further informed by a formative research exploring perspectives of both health service providers and users on use of text based mhealth for supporting self-management in people with type 2 diabetes.
  Arms: Intervention

SUMMARY:
Background: The global prevalence of diabetes is increasing particularly in low and middle income countries like Nepal with the number expected to rise in the near future. Advances in technology have led to greater use of mobile health (mhealth) for managing chronic diseases. mhealth offers a cost-effective way to improve health outcomes with evidence supporting feasibility, acceptability and effectiveness in resource-limited settings like Nepal. However, while mhealth has shown promising results in promoting positive health behaviour and improving service utilization for chronic conditions, its potential for self-management of type 2 diabetes in Nepal is yet to be evaluated. This study thus aims to determine the effectiveness and acceptability of a text based mhealth intervention that improve self-management in people with Type 2 Diabetes in Nepal.

Methods: This study is a 6 month, open-label, two-armed parallel group randomized control trial among 154 participants with type 2 diabetes. Participants will be randomly assigned to either intervention or control group on a 1:1 basis. The intervention group will receive a text based mhealth intervention (text messages) in addition to standard care while the control group will receive only standard care. Baseline data will be collected using a structured questionnaire. Follow up will be done 6 months after the intervention. The primary outcome of the study will be a difference in mean in the HbA1c level from baseline to follow up. The secondary outcomes include changes in diabetes self-care activities, self-efficacy, social-support, diabetes related stress, quality of life and acceptability of the intervention. An economic evaluation will be conducted using a patient perspective. Data will be analyzed using Stata version 13.0.

DETAILED DESCRIPTION:
Background and rationale The number of people living with diabetes has increased globally and is on rapid rise among low and middle income countries (LMICs). In 2021, there were 537 million people living with diabetes and this number is expected to rise to 643 million by 2030 and 783 million by 2045. More than three in four adults with diabetes are living in LMICs. Diabetes accounted for 6.6 million deaths in 2021 and is a major cause of blindness, kidney failure, heart attack, stroke and lower limb amputation. Following the global trend, the prevalence of diabetes has been increasing in Nepal. The International Diabetes Federation (IDF) estimated a prevalence of 8.7% among Nepalese population and the proportion is to rise to 9.4% by 2045.

The burgeoning burden of disease may place serious challenges on the resource constrained national health system due to complications resulting from the disease, coupled with issues around service availability; readiness and limited awareness among the people living with diabetes.

Access to care is of utmost importance for people with diabetes in the course of their disease however, the availability and utilisation of diabetes care services vary across socio-economic and geographical distribution indicating challenges in accessing the diabetes care services. WHO STEPS survey Nepal 2019 reported about three-fourth (73.5%) of the people were not aware of their raised blood sugar. Despite being aware of their condition, about 6% were not on treatment. Similarly, only 70% of adults with raised blood sugar reported compliance to medications to control their blood sugar. In addition, public health facilities in Nepal are not ready to deal with the increasing burden of NCDs including diabetes in terms of qualified health staff, training, availability of equipment and medicines as well as availability of diabetes services in general.

Early diagnosis, treatment and self-management are essential for the prevention and control of the disease. Self-management refers to the activities and behaviour undertaken by the individuals to control and treat their conditions to improve their health outcomes with support from family members, friends and relatives and in consultation with health service providers. The American Association of Diabetes Educators (AADE) has identified seven self-care behaviours for successful and effective self-management of diabetes as healthy coping, healthy eating, being active, taking medication, monitoring, reducing risks and problem solving. Self-management has been proved to be cost effective through reduction in hospital admissions and health care costs. Besides, it is shown to improve HbA1c level and has a positive effect on other clinical, psychosocial, and behavioural aspects of diabetes along with improvement in quality of life by reducing onset and/or advancement of diabetes complications.

With the development of technology, the application of mobile health (mhealth) is becoming increasingly popular in the self-care of chronic diseases. mhealth interventions have been proved to be a therapeutic strategy that could improve the diabetes management despite their economic status. According to the National Population and Housing Census report 2021, about three-fourth (73%) of the households have at least some form of smartphone penetration and 37.9% household with internet access in Nepal.

In the resource limited countries like Nepal, mhealth technology can be a cost-effective approach to deliver care and improve the health outcomes. There are studies demonstrating the feasibility, acceptability and even effectiveness of mhealth in improving the health outcomes for hypertension in Nepal. There is also existing evidence of mhealth as an effective means to communicate health related information and supporting positive behaviour change in a short period of time. Despite availability of body of evidence on acceptability of mhealth in improving service utilization and health outcomes for chronic conditions, the application of behaviour change interventions through mhealth for self-management of diabetes is yet to be evaluated.

Objectives This study aims to determine the effectiveness and acceptability of a text based mhealth intervention that improve self-management in people with Type 2 Diabetes using a co-designed approach in Nepal.

Objective 1: To determine effectiveness and cost effectiveness of text based mhealth intervention in improving self-management (HbA1c level, self-efficacy, perceived support, diabetes related stress, health related quality of life and self-care behaviors) Objective 2: To determine acceptability of a text based mhealth intervention in improving self-management among people with type 2 diabetes

ELIGIBILITY:
Inclusion Criteria:

* adults aged 18 years and above
* clinical diagnosis of type 2 diabetes
* participant who have a mobile phone and is able to read the message on their own or with the help of family members.

Exclusion Criteria:

* not physically or mentally able, not able to provide consent
* pregnant in case of female

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 154 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-25 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c level | six months
  change in mean HbA1c between intervention and control group from baseline to follow up (6 months after the intervention)

CONTACTS AND LOCATIONS:
Locations (1):
- Dhulikhel Hospital, Kavrepalanchowk, Bagmati, Nepal

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ni Z, Atluri N, Shaw RJ, Tan J, Khan K, Merk H, Ge Y, Shrestha S, Shrestha A, Vasudevan L, Karmacharya B, Yan LL. Evaluating the Feasibility and Acceptability of a Mobile Health-Based Female Community Health Volunteer Program for Hypertension Control in Rural Nepal: Cross-Sectional Study. JMIR Mhealth Uhealth. 2020 Mar 9;8(3):e15419. doi: 10.2196/15419. PMID 32149712
- [Background] Bhandari B, Narasimhan P, Jayasuriya R, Vaidya A, Schutte AE. Effectiveness and Acceptability of a Mobile Phone Text Messaging Intervention to Improve Blood Pressure Control (TEXT4BP) among Patients with Hypertension in Nepal: A Feasibility Randomised Controlled Trial. Glob Heart. 2022 Feb 23;17(1):13. doi: 10.5334/gh.1103. eCollection 2022. PMID 35342691
- [Background] Xiong S, Berkhouse H, Schooler M, Pu W, Sun A, Gong E, Yan LL. Effectiveness of mHealth Interventions in Improving Medication Adherence Among People with Hypertension: a Systematic Review. Curr Hypertens Rep. 2018 Aug 7;20(10):86. doi: 10.1007/s11906-018-0886-7. PMID 30088110
- [Background] Wang Y, Min J, Khuri J, Xue H, Xie B, A Kaminsky L, J Cheskin L. Effectiveness of Mobile Health Interventions on Diabetes and Obesity Treatment and Management: Systematic Review of Systematic Reviews. JMIR Mhealth Uhealth. 2020 Apr 28;8(4):e15400. doi: 10.2196/15400. PMID 32343253
- [Background] Lu X, Yang H, Xia X, Lu X, Lin J, Liu F, Gu D. Interactive Mobile Health Intervention and Blood Pressure Management in Adults. Hypertension. 2019 Sep;74(3):697-704. doi: 10.1161/HYPERTENSIONAHA.119.13273. Epub 2019 Jul 22. PMID 31327259
- [Background] Kitsiou S, Pare G, Jaana M, Gerber B. Effectiveness of mHealth interventions for patients with diabetes: An overview of systematic reviews. PLoS One. 2017 Mar 1;12(3):e0173160. doi: 10.1371/journal.pone.0173160. eCollection 2017. PMID 28249025
- [Background] Kang H, Park HA. A Mobile App for Hypertension Management Based on Clinical Practice Guidelines: Development and Deployment. JMIR Mhealth Uhealth. 2016 Feb 2;4(1):e12. doi: 10.2196/mhealth.4966. PMID 26839283
- [Background] Sukartini T, Nursalam N, Pradipta RO, Ubudiyah M. Potential Methods to Improve Self-management in Those with Type 2 Diabetes: A Narrative Review. Int J Endocrinol Metab. 2023 Jan 8;21(1):e119698. doi: 10.5812/ijem-119698. eCollection 2023 Jan. PMID 37038539
- [Background] Panagioti M, Richardson G, Small N, Murray E, Rogers A, Kennedy A, Newman S, Bower P. Self-management support interventions to reduce health care utilisation without compromising outcomes: a systematic review and meta-analysis. BMC Health Serv Res. 2014 Aug 27;14:356. doi: 10.1186/1472-6963-14-356. PMID 25164529
- [Background] American Association of Diabetes Educators. An Effective Model of Diabetes Care and Education: Revising the AADE7 Self-Care Behaviors(R). Diabetes Educ. 2020 Apr;46(2):139-160. doi: 10.1177/0145721719894903. Epub 2020 Jan 12. PMID 31928334
- [Background] Powers MA, Bardsley J, Cypress M, Duker P, Funnell MM, Fischl AH, Maryniuk MD, Siminerio L, Vivian E. Diabetes Self-Management Education and Support in Type 2 Diabetes: A Joint Position Statement of the American Diabetes Association, the American Association of Diabetes Educators, and the Academy of Nutrition and Dietetics. J Acad Nutr Diet. 2015 Aug;115(8):1323-34. doi: 10.1016/j.jand.2015.05.012. Epub 2015 Jun 5. No abstract available. PMID 26054423
- [Background] Adhikari B, Pandey AR, Lamichhane B, Kc SP, Joshi D, Regmi S, Giri S, Baral SC. Readiness of health facilities to provide services related to non-communicable diseases in Nepal: evidence from nationally representative Nepal Health Facility Survey 2021. BMJ Open. 2023 Jul 9;13(7):e072673. doi: 10.1136/bmjopen-2023-072673. PMID 37423630
- [Background] Upreti SR, Lohani GR, Magtymova A, Dixit LP. Strengthening policy and governance to address the growing burden of diabetes in Nepal. WHO South East Asia J Public Health. 2016 Apr;5(1):40-43. doi: 10.4103/2224-3151.206551. PMID 28604396
- [Background] Gyawali B, Ferrario A, van Teijlingen E, Kallestrup P. Challenges in diabetes mellitus type 2 management in Nepal: a literature review. Glob Health Action. 2016 Oct 18;9:31704. doi: 10.3402/gha.v9.31704. eCollection 2016. PMID 27760677
- [Background] Ghimire U, Shrestha N, Adhikari B, Mehata S, Pokharel Y, Mishra SR. Health system's readiness to provide cardiovascular, diabetes and chronic respiratory disease related services in Nepal: analysis using 2015 health facility survey. BMC Public Health. 2020 Jul 25;20(1):1163. doi: 10.1186/s12889-020-09279-z. PMID 32711487
- [Background] Shrestha DB, Budhathoki P, Sedhai YR, Marahatta A, Lamichhane S, Nepal S, Adhikari A, Poudel A, Nepal S, Atreya A. Type 2 Diabetes Mellitus in Nepal from 2000 to 2020: A systematic review and meta-analysis. F1000Res. 2021 Jul 7;10:543. doi: 10.12688/f1000research.53970.2. eCollection 2021. PMID 34621512
- [Background] Dhungana RR, Pandey AR, Shrestha N. Trends in the Prevalence, Awareness, Treatment, and Control of Hypertension in Nepal between 2000 and 2025: A Systematic Review and Meta-Analysis. Int J Hypertens. 2021 Mar 2;2021:6610649. doi: 10.1155/2021/6610649. eCollection 2021. PMID 33747559
- [Derived] Shrestha N, Simkhada P, Kurmi O, Gautam S, Karmacharya B, Shrestha A, Tamrakar R, Poudel AN. Self-management of type 2 diabetes using a co-designed text based mobile health (mHealth) intervention in Nepal: A study protocol for randomised controlled trial. PLoS One. 2025 Nov 4;20(11):e0335333. doi: 10.1371/journal.pone.0335333. eCollection 2025. PMID 41187147
- See also: Related Info — https://www.who.int/news-room/fact-sheets/detail/diabetes
- See also: Related Info — https://www.who.int/docs/default-source/nepal-documents/ncds/ncd-steps-survey-2019-compressed.pdf?sfvrsn=807bc4c6_2
- See also: Related Info — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8719183/
- See also: Related Info — https://censusnepal.cbs.gov.np/results/downloads/national
- See also: Related Info — https://joghep.scholasticahq.com/article/36187-using-mobile-health-to-strengthen-the-communication-skills-for-effective-delivery-of-health-information-in-nepal-a-qualitative-study-of-the-perspecti